CLINICAL TRIAL: NCT04798508
Title: EXPRE-SON-REA : Expressive Versus Neutral Own Names in Neurophysiologic Prognosis Assessment of Intensive Care Unit Comatose Patients.
Brief Title: EXPRE-SON-REA : Expressive Own Names in Neurophysiologic Assessment of Comatose Patients
Acronym: EXPRESONREA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2020-A00747-32
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-01

CONDITIONS: Comatose; Neurophysiologic Abnormality
Keywords: DOC patients; ERP (Event related Potentials); Consciousness
MeSH Terms: conditions — Coma

STUDY DESIGN:
Intervention Model Description: Open and prospective study.
  Evoked related potentials are recorded for each participant while they listen 3 paradigms successively and in a random order:
  i) their own name uttered by a smiling voice ii) their own name uttered by a neutral voice iii) their own name uttered by a rough voice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole group (Other): The whole group listen successively the 3 paradigms :
  * P3 own-name recorded by listening to a smiling voice
  * P3 own-name recorded by listening to a neutral voice
  * P3 own-name recorded by listening to a rough voice
  Interventions: Other: Evoked related potential - P3 paradigm

INTERVENTIONS:
Other: Evoked related potential - P3 paradigm — Evoked related potential are performed for each patient during listen to its own name uttered by i) a neutral voice ii) a smiling voice iii) a rough voice

SUMMARY:
Evaluating the neurologic prognosis in disorders of consciousness (DOC) patients is still a crucial issue in intensive care units.

Neurophysiology allows the investigators to record cerebral responses of patients to auditory stimuli and in particularly to their own name. Numerous studies try to improve the relevance of the auditory stimuli used in this paradigm.

Here the investigators assess if the use of own name stimuli uttered by more expressive voices (for example smiling voices) modulates the cerebral responses recorded. They then correlate these cerebral responses to the neurologic prognosis at three months.

DETAILED DESCRIPTION:
Late auditory evoked potentials (as P3 wave) are used in neurophysiology to assess the level of consciousness in DOC (disorder of consciousness) patients. The P3 wave, elicited by listening standard and deviant stimuli, corresponds to the activation of a frontoparietal network and is considered to reflect a cognitive attention task. Using the own name of the patient as deviant stimuli improve the ability to detect the P3 wave because of the particularly relevance of this stimulus for the patient. However the correlation of this P3 wave and neurologic prognosis is still imperfect and depends on the etiology of the DOC.

In human cognition, to identify the expressivity valence of a voice is essential. Neural processing of expressive voices involves more widespread brain areas than neutral voices processing.

Here the investigators assume that using own name stimuli uttered by more expressive voices (positive : smiling voice or negative : rough voice) should recruit more widespread brain areas and modulate the cerebral responses recorded. The investigators then evaluate if these cerebral responses are relevant markers of consciousness and correlate them to neurologic prognosis at three months.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Disorder of consciousness defined as :

Glasgow coma scale < 8 or >8 but

* eyes opening to pain only
* No response to basic command
* Available neuro-imagery (CT-scan or MRI)
* Normal temperature (no fever or hypothermia)
* Normal blood pressure during neurophysiologic evaluation
* Given consent from relatives

Exclusion Criteria:

* Brain death
* Known deafness
* Severe sepsis uncontrolled during neurophysiologic evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Positive predictive values of P3a responses to own-names uttered by expressive voices (smiling and rough voices) and neutral voices for the neuroprognosis at 3 months | 3 months from DOC evaluation
  Determination of the positive predictive values of the occurence of the P3a wave recorded with expressive and neutral voices for neuroprognostic assessment at 3 months (according to the GOS-E scale)
Negative predictive values of P3a responses to own-names uttered by expressive voices (smiling and rough voices) and neutral voices at 3 months for the neuroprognosis at 3 months | 3 months from DOC evaluation
  Determination of the negative predictive values of the occurence of the P3a wave recorded with expressive and neutral voices for neuroprognostic assessment at 3 months (according to the GOS-E scale)
Sensitivity of P3a responses occurences to own-names uttered by expressive voices (smiling and rough voices) and neutral voices at 3 months for the neuroprognosis at 3 months | 3 months from DOC evaluation
  Determination of the sensibility of the occurence of the P3a wave recorded with expressive and neutral voices for neuroprognostic assessment at 3 months (according to the GOS-E scale)
Specificity of P3a responses to own-names uttered by expressive voices (smiling and rough voices) and neutral voices at 3 months for the neuroprognosis at 3 months | 3 months from DOC evaluation
  Determination of the specificity of the occurence of the P3a wave recorded with expressive and neutral voices for neuroprognostic assessment at 3 months (according to the GOS-E scale)

SECONDARY OUTCOMES:
Negative predictive value of P3a to own-name uttered by expressive voices and neutral voices according to the CRS-r scale | 7, 14 and 28 days from DOC evaluation
  Determination of the negative predictive value of P3a waves (present or absent) for neuroprognostic at 7 days, 14 days and 28 days (according to the CRS-r scale)
Positive predictive value of P3a to own-name uttered by expressive voices and neutral voices according to the CRS-r scale | 7, 14 and 28 days from DOC evaluation
  Determination of the positive predictive value of P3a waves (present or absent) for neuroprognostic at 7 days, 14 days and 28 days (according to the CRS-r scale)
Sensitivity of P3a responses occurences uttered by expressive voices and neutral voices according to the CRS-r scale | 7, 14 and 28 days from DOC evaluation
  Determination of the sensibility of P3a waves (present or absent) for neuroprognostic at 7 days, 14 days and 28 days (according to the CRS-r scale)
Specificity of P3a to own-name uttered by expressive voices and neutral voices according to the CRS-r scale | 7, 14 and 28 days from DOC evaluation
  Determination of the specificity of P3a waves (present or absent) for neuroprognostic at 7 days, 14 days and 28 days (according to the CRS-r scale)
Negative predictive value of P3a to own-name uttered by expressive voices and neutral voices according to eyes-opening | 3 months
  Determination of the negative predictive value of P3a waves (present or absent) for eyes-opening at 3 months
Positive predictive value of P3a to own-name uttered by expressive voices and neutral voices according to eyes-opening | 3 months
  Determination of the positive predictive value of P3a waves (present or absent) for eyes-opening at 3 months
Sensitivity of P3a responses occurences uttered by expressive voices and neutral voices according to eyes-opening | 3 months
  Determination of the sensibility of P3a waves (present or absent) for eyes-opening at 3 months
Specificity of P3a to own-name uttered by expressive voices and neutral voices according to eyes-opening | 3 months
  Determination of the specificity of P3a waves (present or absent) for eyes-opening at 3 months
Description of the amplitudes of the P3a wave to own-name uttered by expressive voices versus neutral voices. | 3 months
  Amplitudes of P3a waves recorded with own name uttered by expressive and neutral voices
Description of the latencies of the P3a wave to own-name uttered by expressive voices versus neutral voices. | 3 months
  Latencies of P3a waves recorded with own name uttered by expressive and neutral voices

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Paris Psychiatrie Neurosciences, Paris, France